CLINICAL TRIAL: NCT00538304
Title: A Study of the Safety and Efficacy of Bimatoprost in Patients With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 192024-035
Record Dates: First submitted 2007-09-28; First posted 2007-10-02 (Estimated); Results first posted 2011-10-27 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): bimatoprost eye drops
  Interventions: Drug: bimatoprost eye drops
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: bimatoprost eye drops — 1 drop in each eye daily for 1 month
  Arms: 1
Drug: placebo — 1 drop in each eye daily for 1 month
  Arms: 2

SUMMARY:
A one month study which will determine the safety and efficacy of bimatoprost eye drops in patients with glaucoma or ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

* Chronic glaucoma or ocular hypertension
* IOP controlled on Xalatan

Exclusion Criteria:

* Uncontrolled medical conditions
* Known hypersensitivity to study medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2007-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Atlanta, Georgia, United States

REFERENCES:
- [Background] Craven ER, Liu CC, Batoosingh A, Schiffman RM, Whitcup SM. A randomized, controlled comparison of macroscopic conjunctival hyperemia in patients treated with bimatoprost 0.01% or vehicle who were previously controlled on latanoprost. Clin Ophthalmol. 2010 Dec 6;4:1433-40. doi: 10.2147/OPTH.S14915. PMID 21188155

RESULTS

PARTICIPANT FLOW:
Groups:
- Bimatoprost Eye Drops: Bimatoprost eye drops
- Placebo: Placebo
Period: Overall Study
Arm/Group | Bimatoprost Eye Drops | Placebo
Started | 151 | 71
Completed | 144 | 66
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost Eye Drops | Placebo | Total
Number analyzed (Participants) | 151 | 71 | 222
Age, Customized [Number; unit: participants]
  < 45 years | 9 | 2 | 11
  Between 45 and 65 years | 66 | 32 | 98
  > 65 years | 76 | 37 | 113
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 44 | 135
  Male | 60 | 27 | 87

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Peak Macroscopic Conjunctival Hyperemia at Month 1
Description: Change from Baseline in macroscopic conjunctival hyperemia (or visible eye redness). Macroscopic conjunctival hyperemia is graded by the investigator who compares the patient's visual appearance of eye redness to standard photographs using a 5-point scale (Scale 0 to +3: none, trace, mild, moderate, severe). The peak change is calculated for each eye by subtracting the largest score across the hourly measurements at baseline from the largest score across the hourly measurements at month 1. A positive number severity grade change from baseline indicated an increase in redness.
Time Frame: Baseline, Month 1
Population: Modified Intent-to-Treat (m-ITT). The m-ITT population included all patients who were enrolled in the study, received at least 1 dose of study medication and were evaluated for macroscopic conjunctival hyperemia at baseline and the month 1 visits.
Measure: Mean (Standard Deviation); unit: Number on a scale (score)
Arm/Group | Bimatoprost Eye Drops | Placebo
Number analyzed (Participants) | 147 | 71
Number on a scale (score)
  Baseline | 0.32 (0.280) | 0.30 (0.288)
  Month 1 | 0.18 (0.456) | 0.02 (0.321)

2. Secondary Outcome: Percentage of Patients With an Increase in Macroscopic Conjunctival Hyperemia in Either Eye at Month 1
Description: Percentage of patients with a >= 1 unit increase in macroscopic conjunctival hyperemia in either eye at the Month 1, 8 AM time point. Macroscopic conjunctival hyperemia is graded by the investigator who compares the patient's visual appearance of eye redness to standard photographs using a 5-point scale (Scale 0 to +3: none, trace, mild, moderate, severe).
Time Frame: Month 1
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Bimatoprost Eye Drops | Placebo
Number analyzed (Participants) | 147 | 71
Percentage of Patients | 8.16 | 1.41

3. Secondary Outcome: Change From Baseline in Mean Intraocular Pressure (IOP) at Month 1
Description: Change from baseline in mean (average) IOP at Month 1 8 AM timepoint. IOP is a measurement of the fluid pressure inside the eye. For each eye, the IOP was either the average of the 2 measurements, or, if a third measurement was required, the median of the 3 measurements. A negative number change from Baseline indicated a reduction in IOP.
Time Frame: Baseline, Month 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Bimatoprost Eye Drops | Placebo
Number analyzed (Participants) | 147 | 71
millimeters of mercury (mmHg)
  Baseline, 8AM | 18.2 (3.13) | 18.0 (3.34)
  Month 1, 8AM | -1.0 (2.64) | 3.6 (3.85)

4. Secondary Outcome: Percentage of Physicians Who Were Very or Extremely Willing to Continue Patient on Drug, if Drug Were Marketed at Month 1
Description: Percentage of physicians who were very or extremely willing to continue patient on drug if drug were marketed based on their reported response to the question. Physicians were asked "Overall, based on how well this drug lowered THIS patient's IOP, balanced with any adverse events she/he may have experienced, would you consider continuing THIS medication (if the drug was marketed)?". The responses were extremely willing, very willing, somewhat willing and not willing. If not willing, physician was asked for reason.
Time Frame: Month 1
Population: as for outcome 1
Measure: Number; unit: Percentage of Physicians
Arm/Group | Bimatoprost Eye Drops | Placebo
Number analyzed (Participants) | 147 | 71
Percentage of Physicians | 85.7 | 39.5

5. Secondary Outcome: Percentage of Patients Who Were Very or Extremely Willing to Use This Glaucoma Medication at Month 1
Description: Percentage of patients who were very or extremely willing to continue to use this glaucoma medication based on their reported response to the question. Patients were asked "Overall, based on how well this drug lowered your IOP, your concern about the preservation of your vision, balanced with any side effects you may have experienced using your medication, would you be willing to continue this medication (eye drops) if your physician prescribed it?". The responses were extremely willing, very willing, somewhat willing and not willing. If not willing, patient was asked for reason.
Time Frame: Month 1
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Bimatoprost Eye Drops | Placebo
Number analyzed (Participants) | 147 | 71
Percentage of Patients | 88.5 | 52.9

6. Secondary Outcome: Percentage of Patients Who Reported No Change in the Appearance of Their Eyes Since the Beginning of the Study at Month 1
Description: Percentage of patients who reported no change in the appearance of their eyes since the beginning of the study. Patients were asked "Are you experiencing a change in how your eye looks now since you began your current glaucoma medication?". The responses were yes or no. If yes, patient was asked for primary reason and if better, worse or as expected based on what the doctor's office told them to expect.
Time Frame: Month 1
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Bimatoprost Eye Drops | Placebo
Number analyzed (Participants) | 147 | 71
Percentage of Patients | 95.1 | 94.1

ADVERSE EVENTS:
Description: The safety population consisted of all patients who were randomized, received at least 1 dose of masked study medication and had at least 1 post-baseline visit.
Arm/Group | Bimatoprost Eye Drops | Placebo
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/71
Other Adverse Events (participants affected / at risk) | 10/150 | 2/71
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost Eye Drops (N=150) | Placebo (N=71)
Conjunctival hyperaemia (Eye disorders) | 10 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo